CLINICAL TRIAL: NCT05751213
Title: Effects of Pelvic Floor Muscle Exercises With and Without Knack Technique in Post-menopausal Women With Stress Urinary Incontinence
Brief Title: Knack Technique in Post-menopausal Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0506
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence,Stress
Keywords: exercise; pelvic floor; post menopause; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- knack technique. (Experimental): pelvic floor muscle exercises with knack technique.
  Interventions: Other: knack technique.; Other: pelvic floor muscle exercises
- pelvic floor muscle exercises (Active Comparator): pelvic floor muscle exercises
  Interventions: Other: pelvic floor muscle exercises

INTERVENTIONS:
Other: knack technique. — It consists of 11 patients who will receive pelvic floor muscle exercise and knack technique at outpatient clinic and at home. 8 maximum voluntary contractions of pelvic floor muscles in supine sustained for 6s with a resting interval twice as long between contractions, followed by 3 fast contractions. 3 times per day. 3 days per week at home for 3 months. 3 exercises in supine position. 8 repetitions of each exercise 3times per day , 3 days per week. .
  Orientation to perform the knack during activities of daily life. The knack consists of voluntary pelvic floor muscles contraction before and during activities that increase abdominal pressure.
  The exercise will be performed in the supine (first month), sitting (second month), and standing (third month) positions twice a month for 3 months at outpatient clinic. (6 outpatient sessions)
  Arms: knack technique.
Other: pelvic floor muscle exercises — It consists of 11 patients who will receive pelvic floor muscle exercises at the outpatient and at home. 8 maximum voluntary contractions of pelvic floor muscles in supine position sustained for 6s with a resting interval twice as long between contractions followed by 3 fast contractions. 3 times per day , 3 days per week at home for 3 months. Two sessions per month at outpatient clinic for 3 months

SUMMARY:
To determine the Effects of pelvic floor muscle exercise with and without Knack Technique in post-menopausal women with stress urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Multiparous women
* Previous history of vaginal deliveries
* Women with mild to moderate stress or mixed incontinence (with predominance of SUI) via the 3 incontinence questions (3IQ)
* Able to have a gynecological examination

Exclusion Criteria:

* Symptoms of overactive bladder alone
* Previous participation in a pelvic floor re-education program and/or previous pelvic floor surgery or currently receiving other treatment for urinary incontinence.
* Loss of stools or mucus
* Active urinary or vaginal infection in the past 3 months

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — post-menopausal women
Enrollment: 22 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
3 DAY BLADDER DIARY | 12th week
  It is a validated instrument which assesses day time and night time urine leakage episodes during consecutive 3 days. IN column indicates how much you drink and when you drink. OUT column indicates how much urine you pass when you go to toilet. Every time you leak put a cross in OUT column. When you go to bed put a line on the chart next to time. This can tell how many times you have to get up to pass urine.

SECONDARY OUTCOMES:
PERFECT SCHEME | 12th week
  The perfect scheme has demonstrated reliability and validity as an assessment tool. Pelvic floor muscles will be assessed by two finger vaginal palpation. The examiner will place fingers at vaginal introitus at about 4cm and the function will be assessed by PERFECT scheme. Modified oxford grading scale (scores of 0-5) will assess the pelvic floor muscle strength.
THE INCONTINENCE QUALITY OF LIFE QUESTIONNAIRE (I-QOL) | 12th week
  The incontinence quality of life questionnaire is a valid instrument for measuring quality of life. The incontinence quality of life questionnaire assesses the impact of stress urinary incontinence on quality of life. The limitations in human behavior, psychosocial impact and social embarrassment is evaluated by I-QOL

CONTACTS AND LOCATIONS:
Overall Officials: hina gul gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Shalamar Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertotto A, Schvartzman R, Uchoa S, Wender MCO. Effect of electromyographic biofeedback as an add-on to pelvic floor muscle exercises on neuromuscular outcomes and quality of life in postmenopausal women with stress urinary incontinence: A randomized controlled trial. Neurourol Urodyn. 2017 Nov;36(8):2142-2147. doi: 10.1002/nau.23258. Epub 2017 May 16. PMID 28508398
- [Background] Bo K. Physiotherapy management of urinary incontinence in females. J Physiother. 2020 Jul;66(3):147-154. doi: 10.1016/j.jphys.2020.06.011. Epub 2020 Jul 21. No abstract available. PMID 32709588
- [Background] Kolodynska G, Zalewski M, Rozek-Piechura K. Urinary incontinence in postmenopausal women - causes, symptoms, treatment. Prz Menopauzalny. 2019 Apr;18(1):46-50. doi: 10.5114/pm.2019.84157. Epub 2019 Apr 9. PMID 31114458
- [Background] Fitz FF, Gimenez MM, de Azevedo Ferreira L, Matias MMP, Bortolini MAT, Castro RA. Effects of voluntary pre-contraction of the pelvic floor muscles (the Knack) on female stress urinary incontinence-a study protocol for a RCT. Trials. 2021 Jul 23;22(1):484. doi: 10.1186/s13063-021-05440-0. PMID 34301324
- [Background] Alves FK, Riccetto C, Adami DB, Marques J, Pereira LC, Palma P, Botelho S. A pelvic floor muscle training program in postmenopausal women: A randomized controlled trial. Maturitas. 2015 Jun;81(2):300-5. doi: 10.1016/j.maturitas.2015.03.006. Epub 2015 Mar 14. PMID 25862491
- [Background] Tosun OC, Solmaz U, Ekin A, Tosun G, Gezer C, Ergenoglu AM, Yeniel AO, Mat E, Malkoc M, Askar N. Assessment of the effect of pelvic floor exercises on pelvic floor muscle strength using ultrasonography in patients with urinary incontinence: a prospective randomized controlled trial. J Phys Ther Sci. 2016 Jan;28(2):360-5. doi: 10.1589/jpts.28.360. Epub 2016 Feb 29. PMID 27065519
- [Background] Tugtepe H, Thomas DT, Ergun R, Kalyoncu A, Kaynak A, Kastarli C, Dagli TE. The effectiveness of transcutaneous electrical neural stimulation therapy in patients with urinary incontinence resistant to initial medical treatment or biofeedback. J Pediatr Urol. 2015 Jun;11(3):137.e1-5. doi: 10.1016/j.jpurol.2014.10.016. Epub 2015 Mar 12. PMID 25824876
- [Background] Yates A. Female pelvic floor 2: assessment and rehabilitation. Nursing Times 2019b. 2019;115(6):30-3
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322